CLINICAL TRIAL: NCT04652037
Title: Visual Outcomes and Rotational Stability of the Acrysof IQ Vivity Toric Extended Vision Intraocular Lens
Brief Title: Visual Results of the Acrysof IQ Vivity Toric Extended Vision Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20.263
Record Dates: First submitted 2020-11-23; First posted 2020-12-03 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Cataract; Presbyopia; Corneal Astigmatism
Keywords: Extended Vision Intraocular Lens; Toric Intraocular Lens; Visual Outcomes; Rotational Stability; Postoperative Visual Disturbances; Patient Satisfaction; Cataract Surgery
MeSH Terms: conditions — Cataract; Presbyopia; Astigmatism; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acrysof IQ Vivity Toric Extended Vision Intraocular Lens Implantation (Experimental)
  Interventions: Device: Acrysof IQ Vivity Toric Extended Vision Intraocular Lens Implantation

INTERVENTIONS:
Device: Acrysof IQ Vivity Toric Extended Vision Intraocular Lens Implantation — Implantation during bilateral cataract surgery of a new non-diffractive extended vision presbyopia and astigmatism correcting intraocular lens (Acrysof IQ Vivity Toric Extended Vision Intraocular Lens)
  Other Names: DFT315, DFT415, or DFT515 Intraocular Lens Implantation

SUMMARY:
The main goal of this study is to evaluate real-world visual outcomes, rotational stability, and patient reported visual disturbances with a non-diffractive extended vision presbyopia and astigmatism correcting intraocular lens in patients with significant corneal astigmatism undergoing bilateral cataract surgery. This is important to ensure optimal results for patients who wish to have intraocular lenses that correct presbyopia and astigmatism, thus giving them a greater independence from spectacles and a better quality of life.

DETAILED DESCRIPTION:
It is estimated that cataracts are the cause of 33% of visual impairment and 51% of total blindness worldwide. Indeed, they are the most important cause of total blindness and preventable blindness in the world. To reduce the burden of this disease, many advances have been made in the field of cataract surgery and have resulted in better visual outcomes. With the development of different types of intraocular lenses over the years, it is now possible to not only treat cataracts, but also tackle presbyopia and astigmatism to increase patients' independence from spectacles and thus improving quality of life. Indeed, the desire for independence from corrective lenses is an important motivation for many patients, which explains the increasingly common use of intraocular lenses correcting for presbyopia.

For most uncomplicated cataract surgeries today in Quebec, Canada, monofocal lens are implanted and their cost is covered by the government. Generally, this lens allows patients to be emmetropic, which translates to good distance vision. However, these patients will need reading glasses for intermediate and near vision. A good proportion of patients are unsatisfied with being dependent on corrective lenses, especially if they did not have any before surgery. There is a correction technique for presbyopia called "monovision", which involves making the patient's dominant eye emmetropic and making the other eye more myopic. This way, the patient can use the myopic eye for intermediate and near vision. Intermediate vision is useful for computer work, for example, while near vision is useful for reading. "Monovision" requires good tolerance of anisometropia by the patient and may interfere with stereoacuity, which may limit its use.

Multifocal intraocular lenses were first implanted in 1986, but took several years to become more commonly adopted. The terms "bifocal" or "trifocal" refer to the number of distinct foci in the lens, allowing the patient to see at different distances. The simultaneous perception of these multiple focal points can be initially disturbing for the patient and may require several months of postoperative neuroadaptation. There are two types of multifocal lenses: refractive and diffractive lenses. Refractive lenses have concentric rings centrifugally increasing in dioptric power on their anterior surface. Diffractive lenses, on the other hand, have diffractive rings on their posterior portion. Meta-analyses have shown that multifocal lenses cause visual disturbances, such as halos and glare, that are more bothersome and frequent than in "monovision". However, multifocal lenses show better rates of independence from spectacles than "monovision". Refractive multifocal lenses, compared to diffractive lenses, tend to produce more glare, halos and higher-order aberrations. However, refractive lenses tend to produce better uncorrected distance visual acuity, while diffractive lenses tend to perform better for near vision.

Finally, extended depth of focus (EDOF) lenses are a newer technology that will be discussed in this study. They have an extended continuous focal point as opposed to the fixed focal points of multifocal lenses, which allows for less superimposition of near and far images compared to multifocal lenses. Theoretical interferometry studies also suggest that EDOF lenses produce better images in between intermediate and near vision. A few comparative studies have shown that EDOF lenses show equal or poorer near visual acuity than diffractive lenses, but have equal or better results for intermediate visual acuity. There are also other newer types of intraocular lenses that, due to their novelty, lack enough data at this time. These include accommodative lenses, postoperative non-invasively adjustable lenses and electronic lenses.

Astigmatism is a refractive error caused by an irregularity in the cornea and/or the crystalline lens that prevents the eye from focusing light evenly on the retina. It causes blurred vision at all distances. It is estimated that almost two-thirds of patients undergoing cataract surgery have preoperative corneal astigmatism between 0.25 and 1.25 diopters. 22% of these patients have astigmatism of 1.50 diopters or more. Toric intraocular lens implantation, first introduced in 1992, is the procedure of choice to correct significant corneal astigmatism (1.00 diopter or greater). For optimal correction of astigmatism with the toric lens, precise alignment of the actual lens axis with the calculated preoperative lens axis of placement is required. This is influenced by several factors, a major one being the rotational stability of the lens. Maximum rotational stability has been observed with hydrophobic acrylic lenses. A prospective study with AcrySof Toric lenses showed significant postoperative rotation of more than 10 degrees in only 1.68% of eyes. In fact, the Acrysof IQ Vivity Toric Extended Vision Intraocular Lens is made with the same AcrySof material, which has shown excellent postoperative rotational stability.

To our knowledge, no study to this day has evaluated the refractive visual outcomes of the Acrysof IQ Vivity Toric Extended Vision Intraocular Lens for the correction of presbyopia and corneal astigmatism. This is believed to be the first study of the Acrysof IQ Vivity Toric Extended Vision Intraocular Lens in Canada. Studying the impact of the Acrysof IQ Vivity Toric Extended Vision Intraocular Lens will provide real-world data on visual acuities after bilateral cataract surgery, intraocular lens rotational stability and subjective assessment of postoperative visual disturbances. This is important to ensure optimal results for patients who wish to have intraocular lenses that correct presbyopia and astigmatism, thus giving them a greater independence from spectacles and a better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing uncomplicated cataract surgery with intraocular lens implantation
* Patients motivated by a greater degree of spectacle independence
* Patients possessing with-the-rule astigmatism of ≥ 0.75 diopters (D) or against-the-rule astigmatism of ≥ 0.50 D
* Patients for whom the Barrett Toric Calculator suggests T3-T5 cylinder power AND 15D-25D spherical power in both eyes
* Ability to provide informed consent;
* Ability to be followed for the entire duration of the study.

Exclusion Criteria:

* Ocular comorbidity that might hamper postoperative visual acuity
* Previous refractive surgery
* Expected post-op visual acuity worse than 20/25 (on Snellen chart)
* Refractive lens exchange
* Irregular corneal astigmatism and keratoconus
* Angle Kappa/chord mu ≥ 0.7
* Higher order corneal aberrations > 0.6 root mean square (RMS) units (to exclude irregular corneas)
* Difficulties comprehending written or spoken French or English language
* Patients with physical or intellectual disability (e.g. Down syndrome, Parkinson's disease; unable to fixate)
* Ocular surface disease
* Axial length > 26mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Binocular uncorrected visual acuities for distance (6 meters), intermediate (66 centimeters), and near (40 centimeters) | 3 months
  Evaluation of visual acuity, measured using the Snellen chart.

SECONDARY OUTCOMES:
Mean absolute intraocular lens rotation (subjective) | 1 day, 1 week, 3 months
  Mean absolute calculation of intraocular lens rotation compared to axis of placement using slit-lamp measurements (in degrees)
Percentage of toric intraocular lenses within 5 degrees of axis of placement | 3 months
  Percentage calculation using the number of intraocular lens that have rotated within less than 5 degrees of axis of placement using slit-lamp measurements
Postoperative residual astigmatism | 3 months
  Measurement of astigmatism using manifest refraction measurements (in diopters)
Monocular best corrected distance visual acuities (at 6 meters), and distance corrected intermediate (66 centimeters) and near (40 centimeters) visual acuities | 3 months
  Evaluation of visual acuity, measured using the Snellen chart, while correcting refractive error for distance vision only.
Mean refractive spherical equivalent | 3 months
  Calculations of mean refractive spherical equivalent based on manifest refraction measurements (in diopters)
Refractive accuracy | 3 months
  Percentage calculation of the number of eyes with an absolute prediction error of 0.50 diopters or less based on manifest refraction measurements (in diopters)
Patient reported visual disturbances | 3 months
  Evaluation of patient reported visual disturbances using a validated questionnaire for visual disturbances (QUVID)

OTHER OUTCOMES:
Mean absolute intraocular lens rotation (objective) | 1 day, 1 week, 3 months
  Mean absolute calculation of intraocular lens rotation compared to axis of placement using measures from the OPD-Scan (in degrees)
Mean absolute prediction error | 3 months
  Mean absolute calculation of prediction error based on manifest refraction measurements (in diopters)

CONTACTS AND LOCATIONS:
Overall Officials: Georges Durr, MD, FRCSC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pascolini D, Mariotti SP. Global estimates of visual impairment: 2010. Br J Ophthalmol. 2012 May;96(5):614-8. doi: 10.1136/bjophthalmol-2011-300539. Epub 2011 Dec 1. PMID 22133988
- [Background] Flaxman SR, Bourne RRA, Resnikoff S, Ackland P, Braithwaite T, Cicinelli MV, Das A, Jonas JB, Keeffe J, Kempen JH, Leasher J, Limburg H, Naidoo K, Pesudovs K, Silvester A, Stevens GA, Tahhan N, Wong TY, Taylor HR; Vision Loss Expert Group of the Global Burden of Disease Study. Global causes of blindness and distance vision impairment 1990-2020: a systematic review and meta-analysis. Lancet Glob Health. 2017 Dec;5(12):e1221-e1234. doi: 10.1016/S2214-109X(17)30393-5. Epub 2017 Oct 11. PMID 29032195
- [Background] Talley-Rostov A. Patient-centered care and refractive cataract surgery. Curr Opin Ophthalmol. 2008 Jan;19(1):5-9. doi: 10.1097/ICU.0b013e3282f2d7a3. PMID 18090889
- [Background] Hawker MJ, Madge SN, Baddeley PA, Perry SR. Refractive expectations of patients having cataract surgery. J Cataract Refract Surg. 2005 Oct;31(10):1970-5. doi: 10.1016/j.jcrs.2005.03.065. PMID 16338569
- [Background] Sieburth R, Chen M. Intraocular lens correction of presbyopia. Taiwan J Ophthalmol. 2019 Jan-Mar;9(1):4-17. doi: 10.4103/tjo.tjo_136_18. PMID 30993062
- [Background] Keates RH, Pearce JL, Schneider RT. Clinical results of the multifocal lens. J Cataract Refract Surg. 1987 Sep;13(5):557-60. doi: 10.1016/s0886-3350(87)80114-1. PMID 3312575
- [Background] Alio JL, Plaza-Puche AB, Fernandez-Buenaga R, Pikkel J, Maldonado M. Multifocal intraocular lenses: An overview. Surv Ophthalmol. 2017 Sep-Oct;62(5):611-634. doi: 10.1016/j.survophthal.2017.03.005. Epub 2017 Mar 31. PMID 28366683
- [Background] de Silva SR, Evans JR, Kirthi V, Ziaei M, Leyland M. Multifocal versus monofocal intraocular lenses after cataract extraction. Cochrane Database Syst Rev. 2016 Dec 12;12(12):CD003169. doi: 10.1002/14651858.CD003169.pub4. PMID 27943250
- [Background] Xu X, Zhu MM, Zou HD. Refractive versus diffractive multifocal intraocular lenses in cataract surgery: a meta-analysis of randomized controlled trials. J Refract Surg. 2014 Sep;30(9):634-44. doi: 10.3928/1081597X-20140814-04. PMID 25250421
- [Background] Dominguez-Vicent A, Esteve-Taboada JJ, Del Aguila-Carrasco AJ, Monsalvez-Romin D, Montes-Mico R. In vitro optical quality comparison of 2 trifocal intraocular lenses and 1 progressive multifocal intraocular lens. J Cataract Refract Surg. 2016 Jan;42(1):138-47. doi: 10.1016/j.jcrs.2015.06.040. PMID 26948789
- [Background] Savini G, Schiano-Lomoriello D, Balducci N, Barboni P. Visual Performance of a New Extended Depth-of-Focus Intraocular Lens Compared to a Distance-Dominant Diffractive Multifocal Intraocular Lens. J Refract Surg. 2018 Apr 1;34(4):228-235. doi: 10.3928/1081597X-20180125-01. PMID 29634837
- [Background] Cochener B, Boutillier G, Lamard M, Auberger-Zagnoli C. A Comparative Evaluation of a New Generation of Diffractive Trifocal and Extended Depth of Focus Intraocular Lenses. J Refract Surg. 2018 Aug 1;34(8):507-514. doi: 10.3928/1081597X-20180530-02. PMID 30089179
- [Background] Ferrer-Blasco T, Montes-Mico R, Peixoto-de-Matos SC, Gonzalez-Meijome JM, Cervino A. Prevalence of corneal astigmatism before cataract surgery. J Cataract Refract Surg. 2009 Jan;35(1):70-5. doi: 10.1016/j.jcrs.2008.09.027. PMID 19101427
- [Background] Shimizu K, Misawa A, Suzuki Y. Toric intraocular lenses: correcting astigmatism while controlling axis shift. J Cataract Refract Surg. 1994 Sep;20(5):523-6. doi: 10.1016/s0886-3350(13)80232-5. PMID 7996408
- [Background] Kaur M, Shaikh F, Falera R, Titiyal JS. Optimizing outcomes with toric intraocular lenses. Indian J Ophthalmol. 2017 Dec;65(12):1301-1313. doi: 10.4103/ijo.IJO_810_17. PMID 29208810
- [Background] Miyake T, Kamiya K, Amano R, Iida Y, Tsunehiro S, Shimizu K. Long-term clinical outcomes of toric intraocular lens implantation in cataract cases with preexisting astigmatism. J Cataract Refract Surg. 2014 Oct;40(10):1654-60. doi: 10.1016/j.jcrs.2014.01.044. Epub 2014 Aug 20. PMID 25149554